CLINICAL TRIAL: NCT01560273
Title: A Multi-Center Prospective Study Evaluation Aspen Spinous Process Fixation System for Use in Posterolateral Fusion (PLF) in Patients With Spondylolisthesis
Brief Title: Aspen Spinous Process Fixation System for Use in PLF in Patients With Spondylolisthesis
Status: Terminated | Type: Observational
Why Stopped: Will answer study question through other research means.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ASP-11-002
Record Dates: First submitted 2012-03-15; First posted 2012-03-22 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aspen Spinous Process Fixation Device: The Aspen device provides supplemental posterior fixation for fusion
  Interventions: Device: Aspen Spinous Process Fixation Device

INTERVENTIONS:
Device: Aspen Spinous Process Fixation Device — The Aspen device will be placed as posterior fixation to Posterolateral Fusion (PLF)

SUMMARY:
The purpose of this clinical investigation is to evaluate the clinical outcomes of subject with spondylolisthesis undergoing posterolateral fusion (PLF) surgery utilizing the Aspen™ Spinous Process Fixation System. The Aspen™ device will be evaluated using Oswestry Disability Index (ODI) improvement and success of fusion.

DETAILED DESCRIPTION:
Evaluate the clinical outcomes of subject with spondylolisthesis undergoing posterolateral fusion (PLF) surgery utilizing the Aspen™ Spinous Process Fixation System. The Aspen™ device will be evaluated using Oswestry Disability Index (ODI) improvement and success of fusion.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and older
* Diagnosis of mild segmental instability on standing radiography lateral film defined as degenerative spondylolisthesis ≤ 4mm in dynamic imaging (i.e., flexion/extension)
* Scheduled for an elective single-level posterior decompression and posterolateral fusion using AspenTM spinous process fixation system
* Oswestry Disability Index (ODI) v 2.1 score >30%
* Failed at least 3 months of conservative care (non-surgical) OR has clinical signs of neurological deterioration
* Signed Informed Consent Form

Exclusion Criteria:

Pre-operative

* Marked degenerative spondylolisthesis (>4mm)
* Lesions requiring surgery involving two levels
* Prior surgery at index level or adjacent level
* Prior spinal fusion surgery
* Isthmic or lytic spondylolisthesis
* Incompetent or missing posterior arch at the affected level (e.g. complete laminectomy, pars defect)
* Requires complete laminectomy at level of surgery
* Facet joints at implant level are absent or fractured
* Vertebral body compromise or acute fracture at implant level
* Body mass Index (BMI) ≥ 35
* Known allergy to titanium
* Osteoporosis: SCORE (Simple Calculated Osteoporosis Risk Estimation) will be used to screen subjects requiring DEXA. Subjects with T-score < -2.5 will be excluded
* Paget's disease, osteomalacia, or any other metabolic bone disease
* Use of medications or any drug known to potentially interfere with bone/soft tissue healing (e.g. chronic systemic steroids)
* Planned use of additional segmental fixation (eg. facet screws, anterior/lateral plating, anchored cages)
* Use of Bone Morphogenetic Protein (BMP)*
* Unlikely to comply with the follow-up evaluation schedule
* In the opinion of the Investigator, Subject has history of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation
* Active participation in a clinical trial of another drug or device
* Active systemic infection or any other health condition that would preclude surgery
* History of invasive malignancy, except if the subject has received treatment and displayed no clinical signs and symptoms for at least five years
* Pregnant or planning to become pregnant during study participation
* Involvement in active litigation related to back problems at the time of screening
* Direct involvement in the execution of this protocol
* Pre-existing conditions that could interfere with the evaluation of outcome measures (e.g. musculoskeletal, neuromuscular, etc.)

Intra-operative Exclusion

* Intra-operative visualization of a > 4mm spondylolisthesis not previously noted radiographically
* Any change in the surgical procedure that violates the inclusion/exclusion criteria. (eg. switching to double level procedure; placing pedicle screws as posterior fixation).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 50 years and older with spondylolisthesis requiring a single level posterolateral decompression and posterolateral fusion
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Absolute change in Oswestry Disability Index (ODI) | baseline to 12 months post-operative

SECONDARY OUTCOMES:
Title: Fusion success | 12 Months post-operative
Change in Visual Analogue Scale (VAS) (pain) | Baseline, 6 weeks, 2 weeks, 3 months, 6 months, 12 months, & 24 months
Neurological status | Baseline, 6 weeks, 3 months, 6 months, 12 months, & 24 months
  motor functions, reflexes, and sensory
Operative parameters (estimate blood loss, surgery time, fluoroscopy time, and length of hospital stay) | Surgical Visit
Pain medication usage | Baseline, surgery, 6 weeks, 3 months, 6 months, 12 months, & 24 months
Change in EQ-5D-3L | Baseline, 6 weeks, 3 months, 6 months, 12 months, & 24 months
Change in Zurich Claudication Questionnaire | Baseline, 12 months & 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shah, Principal Investigator — Goodman Campbell brain and Spine
Locations (5):
- United States (5):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Community Orthopedic Medical Group, Mission Viejo, California
  - Goodman Campbell Brian and Spine, Indianapolis, Indiana
  - Buffalo Spine Surgery, Lockport, New York
  - Pacific Spine Specialists, Tualatin, Oregon

IPD SHARING:
Plan to Share IPD: Undecided